CLINICAL TRIAL: NCT01696695
Title: Program for Assessment of Capecitabine (Xeloda) Based First-line Therapies in Metastatic Colorectal Cancer (AXEL Study)
Brief Title: An Observational Study of First-Line Capecitabine Based Chemotherapy in Participants With Metastatic Colorectal Cancer
Acronym: AXEL
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27791
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Carcinoma (mCRC) Participants: Newly diagnosed mCRC participants, who will receive first line capecitabine based chemotherapy according to effective official Summary of Product Characteristics, will be observed. The choice of therapy is based exclusively on the medical decision of the treating physician before study enrollment. The study protocol does not enforce treatment initiation and also do not specify any treatment regimen.
  Interventions: Drug: Capecitabine; Drug: Chemotherapy

INTERVENTIONS:
Drug: Capecitabine — First line capecitabine based oral tablet treatment in line with the effective Summary of Product Characteristics
  Other Names: Xeloda
Drug: Chemotherapy — First line chemotherapy according to effective official Summary of Product Characteristics. The study protocol does not specify any particular therapy.

SUMMARY:
This observational study will evaluate the efficacy and safety of different capecitabine based chemotherapies, alone or in combination with other therapies, as first line treatment of metastatic colorectal cancer in participants during everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed mCRC who have started first-line capecitabine-based chemotherapy in accordance with the current Hungarian label

Exclusion Criteria:

* History of serious or unexpected reaction to fluoropyrimidine therapy
* Hypersensitivity to the active ingredient of Xeloda or to any of the excipients of the product, or to fluorouracil
* Known dihydropyrimidine dehydrogenase deficiency
* Pregnancy or lactation
* Inadequate bone marrow, hepatic or renal function
* Treatment with sorivudine or its chemical analogues (for example, brivudine)
* If any contraindication for any drug used in the combination treatment schedules is present, the drug in question cannot be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with newly diagnosed colorectal cancer who have started first-line capecitabine based chemotherapy alone or in combination with other therapies.
Sampling Method: Non-Probability Sample
Enrollment: 882 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Hungary (22):
  - Szent Margit Hospital, Budapest
  - Fov.Onk.Peterfy S.Utcai Korh.-Rend.Int es Baleseti Kozp., Budapest
  - Semmelweis Egyetem, II. Belgyógyászati Klinika, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Kenezy Korhaz Rendelointezet, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont, Kecskemét
  - Pest Megyei Flor Korhaz; Oncology, Kistarcsa
  - Borsod-Abauj-Zemplen Megyei Korhaz Es Egyetemi Oktato Korhaz; Onkologiai Osztaly, Miskolc
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Pécsi Tudományegyetem Áok; Onkoterapias Intezet, Pécs
  - Szent Lázár Kórház, Salgótarján
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Tolna Megyei Onkormanyzat Balassa Janos Korhaz, Szekszárd
  - Dr. Bugyi Istvan Korhaz, Szentes
  - Szent Gyorgy Korhaz;Fejer Megyei, Székesfehérvár
  - Vas Megyei Markusovszky Korhaz X; Oncoradiology, Szombathely
  - Szent Borbala Korhaz, Tatabanuya
  - Veszprem Megyei Csolnoky; Ferenc Korhaz, Veszprém
  - Zala megyei Önkormányzat Kórház és Rendelõintézet, Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Colorectal Carcinoma (mCRC) Participants: Newly diagnosed metastatic colorectal carcinoma (mCRC) participants, who received first line capecitabine based chemotherapy according to effective official Summary of Product Characteristics, were observed. The choice of therapy was based on exclusively the medical decision of the treating physician before study enrollment. The study protocol did not enforce treatment initiation and also did not specify any treatment regimen.
Period: Overall Study
Arm/Group | Metastatic Colorectal Carcinoma (mCRC) Participants
Started | 882
Completed | 0
Not Completed | 882
Not completed — Disease progression | 373
Not completed — Death | 29
Not completed — Adverse Event | 74
Not completed — Withdrawal by Subject | 92
Not completed — Lost to Follow-up | 48
Not completed — Other | 74
Not completed — Major Protocol Violation | 192

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all enrolled participants who provided evaluable data for efficacy variables.
Groups:
- mCRC Participants: Newly diagnosed mCRC participants, who received first line capecitabine based chemotherapy according to effective official Summary of Product Characteristics, were observed. The choice of therapy was based on exclusively the medical decision of the treating physician before study enrollment. The study protocol did not enforce treatment initiation and also did not specify any treatment regimen.
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289
  Male | 401

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS)
Description: PFS was assessed using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and is defined as the time from the first dose of indicated treatment to disease progression (PD) or death, whichever occurred first. Participants who did not progress or died while being followed were censored on the date of the last visit. Participants without post-baseline tumor assessments were conservatively censored on the date of first study medication, which is PFS was assigned a value of 1 day. PD: at least 20 percent (%) increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 millimeter (mm); progression of existing non-target lesions; or presence of new lesions. Median PFS was estimated using Kaplan-Meier method.
Time Frame: Baseline until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurred first, evaluated up to Day 1254
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Days | 254 [230 to 279]

2. Primary Outcome: PFS by Therapeutic Regimens
Description: PFS was assessed using RECIST v1.1 and is defined as the time from the first dose of indicated treatment to PD or death, whichever occurred first. Participants who did not progress or died while being followed were censored on the date of the last visit. PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm; progression of existing non-target lesions; or presence of new lesions. Median PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT Population. Here, number (n)= number of participants evaluable for the specified therapeutic regimen.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Days
  Capecitabine monotherapy (n=246) | 194 [176 to 224]
  Capecitabine + bevacizumab (n=25) | 391 [129 to NA] — Only 1-sided confidence interval was planned to be calculated for this regimen.
  Capecitabine + irinotecan (n=106) | 242 [177 to 276]
  Capecitabine + irinotecan + bevacizumab (n= 91) | 392 [316 to 525]
  Capecitabine + oxaliplatin (n=173) | 240 [206 to 291]
  Capecitabine + oxaliplatin + bevacizumab (n= 49) | 392 [210 to 442]

3. Secondary Outcome: Percentage of Participants With Overall Response as Assessed by Investigator Using RECIST v1.1
Description: Overall response is defined as a complete response (CR) or a partial response (PR) as determined by the Investigator using RECIST v1.1 on 2 consecutive occasions at least 6 weeks apart. Participants were evaluated for tumor response per RECIST v1.1 and assessed by computed tomography (CT) or magnetic resonance imaging (MRI):CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than (<) 10 mm). No new lesions.PR was defined as greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: as for outcome 1
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Percentage of participants | 24.3 [21.2 to 27.7]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit as Assessed Using RECIST v1.1
Description: Clinical benefit was defined as having a confirmed CR, PR or stable disease (SD) for at least 24 weeks on study according to RECIST v1.1.CR: complete disappearance of all target lesions and non-target disease,with the exception of nodal disease.All nodes,both target and non-target, must decrease to normal (short axis <10 mm).No new lesions.PR: >=30% decrease under baseline of the sum of diameters of all target lesions.The short axis was used in the sum for target nodes,while the longest diameter was used in the sum for all other target lesions.No unequivocal progression of non-target disease.No new lesions.SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,taking as reference the smallest sum diameters while on study.PD:at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions,or presence of new lesions.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Percentage of participants | 82.9 [79.9 to 85.6]

5. Secondary Outcome: Percentage of Participants Who Underwent Metastasectomy
Description: Metastasectomy is the surgical removal of metastases, which are secondary cancerous growths that have spread from cancer originating in another organ in the body.
Time Frame: Baseline up to 1254 days
Population: ITT Population. Here, N (number of participants analyzed) indicates the total number of participants who provided evaluable data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 663
Percentage of participants | 6.2 [4.4 to 8.0]

6. Secondary Outcome: Mean Duration of Capecitabine Therapy
Time Frame: Baseline up to 1254 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | mCRC Participants
Number analyzed (Participants) | 660
Days | 188.8 (171.71)

7. Secondary Outcome: Percentage of Participants With Dose Modification of Capecitabine
Time Frame: Baseline up to 1254 days
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 690
Percentage of participants | 85.6

ADVERSE EVENTS:
Time Frame: Baseline up to Day 1254
Description: Safety Population included all enrolled participants.
Arm/Group | mCRC Participants
Serious Adverse Events (participants affected / at risk) | 55/882
Other Adverse Events (participants affected / at risk) | 140/882
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mCRC Participants (N=882)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 2
Heart failure (Cardiac disorders) | 3
Cardiopulmonary failure (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Large intestine perforatio (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Death (General disorders) | 1
General physical health deterioration (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
White blood cell count decreased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Aphasia (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndroma (Skin and subcutaneous tissue disorders) | 2
Nephrostomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mCRC Participants (N=882)
Diarrhea (Gastrointestinal disorders) | 98
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.